CLINICAL TRIAL: NCT03684161
Title: Cardiopulmonary Function in Adults Born With a Ventricular Septal Defect
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: FEMM4
Record Dates: First submitted 2018-09-06; First posted 2018-09-25 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2018-09

CONDITIONS: Ventricular Septal Defect
Keywords: Congenital Heart Disease; Ventricular Septal Defect; Long-term Outcome; Cardiopulmonary Function
MeSH Terms: conditions — Heart Septal Defects, Ventricular; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Surgically closed VSDs: Patients born with a ventricular septal defect, which have been closed in early childhood.
  Interventions: Diagnostic Test: Cardiopulmonary function
- Small, persistent VSDs: Patients born with a small, hemodynamically insignificant ventricular septal defect.
  Interventions: Diagnostic Test: Cardiopulmonary function
- Healthy controls: Healthy control subjects.
  Interventions: Diagnostic Test: Cardiopulmonary function

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary function — Body composition measurements; Pulmonary function tests; Cardiopulmonary exercise test; Force frequency releationship, ultrasound

SUMMARY:
The overall objective for this study is to evaluate the cardiopulmonary function of VSD-patients compared with healthy age- and gender-matched controls. VSD patients with a surgically corrected defect and VSD patients with a small persistent defect will be included.

DETAILED DESCRIPTION:
1. Title Cardiopulmonary capacity past the age of 40 - adults with either a persistent or a surgically repaired ventricular septal defect
2. Background:

   Over the last decades, the treatment possibilities in pediatric cardiology and cardiac surgery have improved markedly and accordingly, more than 90% of children born with a congenital heart disease now reach adulthood [1,2]. As a result, the population of adults is today greater than that of children with congenital cardiac defects [3] and consequently, the focus has started to shift more towards the long-term outcome of the growing adult population. Among the most common cardiac defects is the ventricular septal defect (VSD), seen as a hole of varying position, size and significance in the wall separating the two pumping chambers of the heart. The VSD occurs at a rate of 2-3 per 1000 life-births [4,5] and is at large diagnosed during childhood. In the first decade of life, approximately 30% of the VSDs will close spontaneously[6], with a declining number closing naturally with increasing age[7]. VSDs that do not close spontaneously are considered to be of either hemodynamic importance or not. Patients born with a hemodynamically significant and operable VSD will undergo surgical or catheter-based closure, mostly at an early age, whereas the rest are considered too small and insignificant to be of any hemodynamic importance.

   Common for both the surgically closed and the small, unrepaired VSDs is that the long-term outcome of these patients is thought to be excellent. Patients who have undergone closure of their defect are considered to be "cured" and few years following successful surgery, they are discharged from further follow-up visits in the health care system. Similarly, patients with small, unrepaired VSDs are followed in their first decades of life with follow-up visits, with the majority being discharged when they reach adulthood. Therefore, very little is known on the possible consequences of a congenital VSD on the physical functioning in later adulthood. Recently, researchers from our institution assessed the physical capacity in both open and closed VSDs, focusing on the early adulthood, and found a number of physical parameters affected in patients when comparing them with their healthy peers. In patients in their early twenties with an operated VSD, a 20% lower exercise capacity and an abnormal contractility was found during physical activity compared with a group of healthy controls [8,9]. Young adults, in their mid-twenties, with small, open VSDs exhibited a similarly reduced exercise capacity as compared with healthy peers [10,11], and in both open and closed patients, health-related quality of life was found to be affected with a lower self-assessed physical functioning compared with healthy controls [9,10].

   Young adults with open and closed VSDs also demonstrated a reduced ventilatory response during exercise [10,12]. This led to further detailed examination of their pulmonary function in a newly completed study on similarly aged patients with either open or closed VSDs[13]. Both patient groups displayed a degree of limited pulmonary function, especially in the dynamic measurements and most pronounced in the surgically corrected patients. Other recent studies have also found degrees of limitations in these patients [14-16]. However, common for all studies is that the patients investigated are usually in their mid-twenties with no patient reaching the age of 40 years. Therefore, it is not yet known whether any of these documented limitations will progress, decrease or stay unchanged with increasing age. As the group of patients with congenital VSDs grows older, age-related factors such as acquired hypertension, coronary artery disease, and other cardiovascular problems will start emerging and perhaps accelerate any former trivial symptoms related to their underlying cardiac anomaly. How this will further affect the already found limitations in young adults is unknown. Therefore, we feel there is an unmet need for a prospective, clinical study investigating how these patients are doing past the age of 40 as compared with their peers.
3. Study objectives and purpose:

   3.1 Objectives: The overall objective of this study is to investigate a group of adults, age 40 or above, who are living with a small, unrepaired or a surgically corrected ventricular septal defect. Outcomes will be illustrated through an extensive pulmonary function study performed at rest, questionnaires, two different exercise studies and a study on heart rate variability through Holter monitor. Results of the two patient groups will be compared with those of healthy, age-matched controls.

   3.2 Hypotheses: I. Adult patients, age 40 or above, with small, unrepaired VSDs or surgically corrected VSDs will demonstrate a reduced pulmonary function at rest compared with healthy, age-matched controls.

   II. Adult patients, age 40 or above, with small, unrepaired VSDs or surgically corrected VSDs will experience a 20% reduced exercise capacity during bicycle exercise tests compared with healthy, age-matched controls.

   III. Adult patients, age 40 or above, with small, unrepaired VSDs or surgically corrected VSDs will experience reduced minute ventilation during bicycle exercise tests compared with healthy, age-matched controls.

   IV. Adult patients, age 40 or above, with small, unrepaired VSDs or surgically corrected VSDs will reach lower scores on health-related quality of life as compared with healthy, age-matched controls.

   V. Adult patients, age 40 or above, with small, unrepaired VSDs or surgically corrected VSDs will reach a maximum of force frequency quicker than healthy, age-matched controls when examined by echocardiography during exercise.

   VI. Adult patients, age 40 or above, with small, unrepaired VSDs or surgically corrected VSDs will have an increased rate of arrhythmias and a reduced heart rate variability compared with healthy controls

   3.2 Endpoints: The primary endpoint of the study is peak oxygen uptake (ml O2/kg/min) during exercise. Secondary endpoints include forced expiratory volume in one second at rest, peak isovolumetric acceleration (cm/s2) during exercise, airway resistance (R5-20), diffusion capacity (DLCO), alveolar volume, health-related quality of life and heart rate.
4. Materials and Methods:

   4.1 Study population: The study population will consist of three groups; a group of small unrepaired VSDs, a group of surgically corrected VSDs and a group of healthy, age-matched controls. Each group is aimed at including 20 participants.

   4.1.1 Inclusion criteria: By searching the Electronic Patient Journal (EPJ), patients born between 1938 and 1978 will be included if they are registered with DX Q21.0; the International Classification of Diseases (ICD) code for a ventricular septal defect, and if the defect is unrepaired in accordance with criteria from the European Society of Cardiology Guidelines [5] or is repaired as documented by the procedural code KFHB. Recruitment of healthy control subjects will take place by means of adverts at the website www.forsoegspersoner.dk. Control subjects will be matched by likewise age-groups.

   4.1.2 Exclusion criteria: Patients and control subjects will be excluded from the project if they meet any one of the following: lack of medical record, serious congenital cardiac abnormalities, lack of Danish language skills, severe lung or heart disease, syndromes, such as Down's, mentally or physically incompetent to perform the bicycle test. Participants will be informed of the exclusion criteria at the initial information interview before inclusion in the study. Oral verification is considered sufficient to verify the exclusion criteria.

   4.1.3 Enrolment: Patients who meet the abovementioned criteria, and control subjects, who show interest will receive a letter. This will include written participation information as well as the appendix "Forsøgspersoners rettigheder i et sundhedsvidenskabeligt forskningsprojekt" and "Før du beslutter dig" composed by the Danish Research Ethics Committee. Through our written information, we urge participants to carefully read this appendix. In the written information the right to bring another person to the meeting is also stated. A reply card and a prepaid envelop will also be included in the letter, with which participants can accept or reject further information of the project. Participants, who accept partaking in the project, will receive a date by their preferred means of contact; telephone, e-mail or a letter. At this date they will meet at the hospital in order to receive oral information on the project. One of the project organisers will furthermore certify that the participant fulfil in- and exclusion criteria. After this, they will be provided with the consent form. The oral session will be allocated as much time as needed for a complete briefing and answering questions and no interference will occur.

   At all times, it will be possible to obtain further information by contacting the project organiser, Marie Maagaard Sørensen or Filip C.A. Eckerström. Contact information will be evident on all material received. Documented travel expenses in connection with participation in the project will be economically reimbursed. Potential project participants will be informed of this through the information material.

   4.2 Study-design: The study is designed as a prospective, long-term follow-up study and will be conducted between September 2018 and June 2021. It consists of five elements; pulmonary function tests performed at rest, a maximal exercise test measuring the peak oxygen uptake of the participant, two questionnaires (one on health-related quality of life, one on habitual physical activity), a supine bicycle test combined with echocardiography for the assessment of cardiac contractility and wearing a Holter monitor. All tests are performed once at the same location.

   The timeframe for the tests are estimated at lasting three hours in total. The order of tests will commence with the assessment of pulmonary function at rest which is estimated at lasting half an hour. After this, the maximal bicycle test measuring oxygen uptake will take place, lasting another half hour. This will be followed by an hour of resting in order to ensure some physical restitution before the supine bicycle test, which is likewise estimated at half an hour. In the hour between the two bicycle tests, the two questionnaires are intended to be completed. Following the second bicycle test, the participant will be equipped with a Holter monitor and will then have completed the full list of examinations. Further details on each test will be mentioned under section 4.5 Data collection.

   4.3 Power calculation: The number of participants needed to be included in order to increase the probability of statistical significance is estimated based on the primary endpoint from Hypothesis I; peak Oxygen uptake during exercise. This has been chosen as a variable as it has previously been found to be statistically and clinically different in young adults with either unrepaired VSDs [10] or surgically corrected VSDs [9] compared with healthy peers. The results from Heiberg et al are chosen for the power calculation, where a reduced peak Oxygen uptake in surgically corrected VSDs of 38.0±8.2) ml O2/kg/min was measured along with a mean value of 47.9‡6.5ml O2/kg/min in healthy, age- and gender-matched controls. It is equally expected in this project that the older patients, both small unrepaired and surgically corrected VSDs, will reach a lower peak Oxygen uptake compared with a healthy group of controls during bicycle exercise. A difference of 80% is likewise expected like that of the previously found difference with the same standard deviations. A statistical power of 90% and a signiﬁcance level of 5% are set, indicating that at least 19 participants are needed to be included in each group. This is considered possible from an assessment of participants fulfilling the inclusion criteria from a diagnosis-code-search in the EPJ-system, where several hundred participants were readily identified. We aim at including 20 participants in each group.

   4.4 Data analyses and statistics All calculations will be carried out using the statistical software Stata 11.2 (StataCorp LP, College Station, TX, USA). For all graphical description, Graph Pad Prism 6 (GraphPad Software, La Jolla, CA, USA) will be used. Continuous, normally distributed data will be reported as means with ±standard deviations (SD) or as medians with 95% confidence intervals or total range. For normally distributed data, the unpaired Student's t-test will be used, and for normally distributed data with unequal SD the unequal Student's t-test will be used. For non-normally distributed data the Mann-Whitney-Wilcoxon rank-sum test will be chosen. Regarding the assessment of reproducibility, which will be relevant when analysis data from Hypothesis V - Contractility during exercise, the Intraclass Correlation Coefﬁcient (ICC)17 will be chosen using a two-way mixed model for the differences between measurements to estimate agreements of inter- and intraobservers. Correlation will be checked using simple regression analyses. A p-value <0.05 will be considered statistically significant for all results.

   4.5 Data collection - test description 4.5.1 Hypothesis I - Pulmonary function at rest In order to thoroughly evaluate the pulmonary function at rest, a number of tests will be applied so the entire ventilatory system will be assessed. Below, each specific lung function test will be considered.

   4.5.1.1 Dynamic lung function The dynamic lung function will be evaluated using a spirometry performed with the Jaeger MasterScreen Pneumo spirometer by Carefusion or the Jager MasterScreen PFTpro diffusion system with bodybox by Intramedic. The tests will be performed in accordance to American Thoracic Society/European Respiratory Society Guidelines [18]. The participants will exhale trough a mouthpiece and the equipment will then be able to measure airway flow dynamics. The test will include forced expiratory volume in one second, forced vital capacity, the ratio between the two volumes, and peak expiratory flow. The values are automatically given by the trial equipment after testing and they will be described as volumes and as percentage of expected.

   4.5.1.2. Plethysmography (Static lung function) The plethysmography will be performed with Intramedics Jaeger MasterScreen PFTpro difussionssystem and Bodybox from CareFusion. The participant sits inside an airtight cabinet where they will ventilate through a single mouthpiece. At the end of normal expiration, the mouthpiece will close and the participant is then asked to make an inspiratory effort. The lungs expand, decreasing pressure within the lungs, increasing lung volume. This in turn increases pressure in the cabinet, and increases bodybox volume. The equipment can then determine different lung parametres of which we will measure total lung capacity, residual volume, functional residual capcity and specific airway resistance (sRAW, kPa/sec) [19].

   4.5.1.3 Lung Clearance Index (LCI) The LCI will be performed using the Ecomedics Exhalyzer D with N2 option for washout, Multiple Breath Washout (MBW) and Single Breath Washout (SBW), by Intramedic. A flowmeter and gas sampling port is fitted to a mouthpiece and connected to a flow-past tube which supply tracer gas during wash-in and remove at the start of washout. With MBW the participant breath trough a mouthpiece and the equipment will trace the wash-out of the tracer gas. The tracer gas will be NO2 which is normally resident in the lungs and neither absorbed nor excreted by the body in any significant degree. NO2 wash-out will be traced during normal tidal ventilation with 100% oxygen and with every breath there should be a gradual fall in peak concentration of the tracer. Wash-out is deemed complete when the end-tidal tracer gas concentration is 1/40th of starting concentration [20-22]. Hereby the equipment can analyse LCI 2,5 (LCI is defined as the cumulative expired volume (CEV) divided by the functional residual capacity (FRC), Scond (ventilation heterogeneity generated in the conductive lung zone) and Sacin (ventilation heterogeneity generated peripheral to the acinar entrance). The values are automatically given by the trial equipment after testing. All values are described as percentage of expected.

   4.5.1.4 Diffusion Capacity: The diffusion capacity test will be performed on the same equipment as the plethysmography. The test determines lung Carbon Monoxide diffusion capacity (DLCO) and alveolar volume (VA) expressed as percentage of expected value. For the DLCO, the participants will ventilate through the mouthpiece. First they will take a deep breath in and exhale to residual volume. Afterwards they will inhale rapidly with a gas mixture containing approximately 0.3% CO, 10% He, 21% O2 and balanced N2. They will hold their breaths for 9 seconds and then exhale rapidly. VA is the volume of distributed helium, expressed in body temperature and pressure saturated (BTPS) units, from a single-breath DLCO test [23]. The values are automatically given by the study equipment after testing.

   4.5.1.5 Impulse Oscillometry (IOS) IOS will be performed using the Carefusion m Vyntus Impulse oscillometer with SentrySuite software and Vyntus Spirometer. Participants will perform normal tidal ventilation through the equipment mouthpiece while the loudspeaker generates an impulse-shaped pressure signal into their respiratory system. They will breath tidally for 30 seconds, as instructed by our trained personal. The equipment will then be able to analyse resistance in of the respiratory system at 5 Hz (R5), and at 20 Hz (R20) and the difference between the two measured resistances (Diff 5-20) [24,25]. It will be ascertained that each test results in at least three reproducible manoeuvres without artifacts caused by coughing, swallowing, vocalization or breath holding. The participants mean values will then be used for further trial analysis. The values are automatically given by the trial equipment after testing.

   4.5.3 Hypothesis II and III - Exercise capacity Exercise capacity will be tested on a Lode Corival ® ergometer cycle. With the Jaeger MaesterScreen CPX software system, we will monitor pulmonary ventilation and gas exchange in a breath-by-breath measurement. During test sessions, heart rate, blood pressure and electrocardiogram, will be measured continuously. An individual workload protocol based on the subject's body-mass, gender and exercise habits will be determined before the first test. Participants are initially examined at rest while strapped on to the ergometer cycle pedals for 2 minutes. Afterwards, they will perform continuous leg exercise with gradually incremented workloads until complete exhaustion. The participants will be instructed to maintain a cycling speed of 60 to 70 rounds/min, not to talk or stand up in the pedals during testing, and to keep pedalling until complete exhaustion. Maximal exhaustion is defined as a respiratory exchange ratio of 1.10 and a heart rate plateau or a plateau of oxygen uptake [26]. Blood pressure will be measured with an arm cuff at every third minute.The assumed test time is 8 to 12 minutes per test.

   4.5.4 Hypothesis IV - Questionnaires Participants will be asked to fill out a questionnaire in order to gather information of the weekly amount of physical activity. This is reviewed with the purpose of illustrating if the patients are restricted in any ways compared to the healthy controls in regards to their exercising habits, and for this assessment, the standardized International Physical Activity Questionnaire (IPAQ) [27] will be chosen. Also, participants will be asked to fill out the health survey Short-Form-36 (SF-36) with the aim of documenting Health-Related-Quality-of-Life (HRQoL). The latter is chosen based on the need for a generalized quality of health questionnaire, which is widely used and thus, provides data which is easily comparable to other studies.

   4.5.5 Hypothesis V - Contractility during exercise Each individual will undergo echocardiographic scans in accordance with recommendations from Dansk Cardiologisk Selskab [28]. Echocardiography will be performed with the participants in supine position, while connected to a bicycle ergometer, in order to carry out an exercise stress echocardiography. Participants will initially be scanned at rest and then start pedalling at a steady pace of app. 60-70 rpm with scans being performed at predefined times with a duration of app. 30 seconds. The test will end with either exhaustion despite encouragement to continue or when a target heart rate of app 160-min is reached (which is measured continuously throughout the test). This target heart rate is chosen as echocardiographic recordings lose quality beyond this level due to heart movements and lung interference [29]. The exercise stress echocardiography is performed in order to gather information on the force-frequency relationship (FFR), which describes the property of the cardiac muscle to change contractile force in accordance with heart rate. Changes in the configuration of the myocardium may alter this ability and result in a sloping of the FFR in patients with cardiac abnormalities compared to healthy subjects [30]. An important measure of FFR is the isolvolumetric acceleration, measured in cm/sec2, as this is not dependent on loading conditions of the pumping chambers, and holds a high rate of reproducibility. It is especially stable in the face of a changing afterload, as it is measured in the isovolumetric contraction period prior to semilunar valve opening.

   4.5.6 Hypothesis VI - Heart rate variability Following the second bicycle test, participants will be equipped with a Holter monitor in order to assess their heart-rate-variability and possible arrhythmias. ECG will be monitored with a 2-channel Holter monitor (SPACELABS HEALTHCARE Lifecard CF Digital Holter Recorder). It will be attached to the subject by the investigators, as instructed by a Holter-Nurse from the Dept. of Cardiology, Aarhus University Hospital. Participants will be instructed in how to handle the Holter monitors at home and provided with an information document on how to handle the Holter monitor and how to return it. They will also be given an incident journal, where they can register if they experience any symptoms they might relate to their cardiopulmonary function, with time of incident. This will be used for the Holter data analysis. Participants will be wearing the Holter monitor for a full 24 hours after activation following the second bicycle test. They will receive a pre-paid addressed return-box and instruction to mail the Holter monitor, memory card, wires, and leftover electrodes back to our institution as soon as the Holter-recording is over. If the Holter monitor is not returned within the first week, we hold the right to contact the participant and remind them to return the Holter monitor until it is in our custody.
5. Ethical Consideration:

   All data will be made anonymous and all included participant will receive a 4-digit identification code which will be evident on all subject study data. The identification list with participant personal data will be stored in REDCap, the legal base of the university. Data for each participant will be stored in their REDcap file (marked with study number). All digitalised data will be stored on two external harddrives that is kept safe behind two locked doors. The study is conducted in accordance with the Helsinki declaration and Danish law. The project will obtain permission from the Danish Protection Agency and the National Committee on Health Research Ethics. Data will be handled in agreement with the personal data handling law and the participants' safety is always the number one priority during this study.

   All examinations throughout this project are free of any risks to the participants. The momentary strain from participating in the tests is judged as being acceptable in the light of the importance this project could have for patients with small, unrepaired or surgically corrected VSDs. The participant safety is always the leading priority of the investigations. Compensations to cover transport expenses will be provided, but not reimbursement to cover lost earnings or any type of payment for participating. This project holds no dependence - neither economically nor in ways of interest - to any potential sponsors. Granted money from foundations will be transferred to a foundation-account which is managed by the Foundation-administration at Aarhus University-hospital, Skejby. Names on potential sponsors will be depicted in later published material.
6. Resources:

   The study is based from the department of Cardiothoracic Surgery on Aarhus University Hospital, which has a longstanding tradition for clinical trials. All tests will be performed by medical personnel who are trained in conduction of clinical studies.The Project Coordinators Marie Maagaard Sørensen and Filip C. A. Eckerstöm have both previously conducted and completed clinical studies at the department. Both are instructed and educated in the trial investigations and will assist the participants during the trial days. They will furthermore function as contacts for the trial. Professor of cardiothoracic surgery Vibeke Elisabeth Hjortdal has vast experience of both clinical and experimental cardiovascular research and will be the main supervisor of the project. All necessary equipment and facilities required to carry out this study are available or provided by the Department of Cardiothoracic and Vascular Surgery, the Department of Paediatrics and the Department of Cardiology at Aarhus University Hospital.
7. Prospective publication:

The project is planned to result in at least one scientific article on the exercise capacity, cardiac contractility, heart rate variability and extended pulmonary function in adults, age 40 or above with a congenital VSD, published in an international journal. Positive as well as negative and inconclusive results will be published.

ELIGIBILITY:
Inclusion:

* Patients born between 1938 and 1978.
* Patients registered with DX Q21.0, and if the defect is unrepaired in accordance with criteria from the ESC guidelines 5 or is repaired as documented by the procedural code KFHB.

Recruitment of healthy control subjects will take place by means of adverts at the website www.forsoegspersoner.dk. Control subjects will be matched by likewise age-groups.

Exclusion:

* Lack of medical record
* Serious congenital cardiac abnormalities
* Lack of Danish language skills
* Severe lung or heart disease
* Syndromes, such as Down's
* Mentally or physically incompetent to perform the tests.

Participants will be informed of the exclusion criteria at the initial information interview before inclusion in the study. Oral verification is considered sufficient to verify the exclusion criteria.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of three groups; a group of small unrepaired VSDs, a group of surgically corrected VSDs and a group of healthy, age-matched controls. Each group is aimed at including 20 participants.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake | One week.
  (ml O2/kg/min)

SECONDARY OUTCOMES:
Forced expiratory volume in one second (FEV1) | One week.
  (L)
Peak isovolumetric acceleration during exercise | One year.
  (cm/s2)
Airway resistance | One week.
  (x)
Diffusion capacity for carbon monoxide | One week.
  (x)
Health-related quality of life | Post hoc evaluation. 1 year.
  (Questionnaire)
Peak heart rate during exercise | One week.
  (beats/min)

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke E Hjortdal, MD, PhD, DMSc, Principal Investigator — Dept. of Cardiothoracic and Vascular Surgery
Locations (1):
- Department of Cardiothoracic and Vascular Surgery, Aarhus C, Denmark

REFERENCES:
- [Background] Larsen SH, Olsen M, Emmertsen K, Hjortdal VE. Interventional Treatment of Patients With Congenital Heart Disease: Nationwide Danish Experience Over 39 Years. J Am Coll Cardiol. 2017 Jun 6;69(22):2725-2732. doi: 10.1016/j.jacc.2017.03.587. PMID 28571637
- [Background] Warnes CA, Liberthson R, Danielson GK, Dore A, Harris L, Hoffman JI, Somerville J, Williams RG, Webb GD. Task force 1: the changing profile of congenital heart disease in adult life. J Am Coll Cardiol. 2001 Apr;37(5):1170-5. doi: 10.1016/s0735-1097(01)01272-4. No abstract available. PMID 11300418
- [Background] Webb GD. Care of adults with congenital heart disease--a challenge for the new millennium. Thorac Cardiovasc Surg. 2001 Feb;49(1):30-4. doi: 10.1055/s-2001-9918. PMID 11243519
- [Background] Warnes CA, Williams RG, Bashore TM, Child JS, Connolly HM, Dearani JA, del Nido P, Fasules JW, Graham TP Jr, Hijazi ZM, Hunt SA, King ME, Landzberg MJ, Miner PD, Radford MJ, Walsh EP, Webb GD. ACC/AHA 2008 Guidelines for the Management of Adults with Congenital Heart Disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (writing committee to develop guidelines on the management of adults with congenital heart disease). Circulation. 2008 Dec 2;118(23):e714-833. doi: 10.1161/CIRCULATIONAHA.108.190690. Epub 2008 Nov 7. No abstract available. PMID 18997169
- [Background] Baumgartner H, Bonhoeffer P, De Groot NM, de Haan F, Deanfield JE, Galie N, Gatzoulis MA, Gohlke-Baerwolf C, Kaemmerer H, Kilner P, Meijboom F, Mulder BJ, Oechslin E, Oliver JM, Serraf A, Szatmari A, Thaulow E, Vouhe PR, Walma E; Task Force on the Management of Grown-up Congenital Heart Disease of the European Society of Cardiology (ESC); Association for European Paediatric Cardiology (AEPC); ESC Committee for Practice Guidelines (CPG). ESC Guidelines for the management of grown-up congenital heart disease (new version 2010). Eur Heart J. 2010 Dec;31(23):2915-57. doi: 10.1093/eurheartj/ehq249. Epub 2010 Aug 27. No abstract available. PMID 20801927
- [Background] Onat T, Ahunbay G, Batmaz G, Celebi A. The natural course of isolated ventricular septal defect during adolescence. Pediatr Cardiol. 1998 May-Jun;19(3):230-4. doi: 10.1007/s002469900291. PMID 9568219
- [Background] Neumayer U, Stone S, Somerville J. Small ventricular septal defects in adults. Eur Heart J. 1998 Oct;19(10):1573-82. doi: 10.1053/euhj.1998.1083. PMID 9820997
- [Background] Heiberg J, Schmidt MR, Redington A, Hjortdal VE. Disrupted right ventricular force-frequency relationships in adults operated for ventricular septal defect as toddlers: abnormal peak force predicts peak oxygen uptake during exercise. Int J Cardiol. 2014 Dec 20;177(3):918-24. doi: 10.1016/j.ijcard.2014.10.009. Epub 2014 Oct 28. PMID 25456699
- [Background] Heiberg J, Laustsen S, Petersen AK, Hjortdal VE. Reduced long-term exercise capacity in young adults operated for ventricular septal defect. Cardiol Young. 2015 Feb;25(2):281-7. doi: 10.1017/S1047951113002084. Epub 2013 Nov 21. PMID 24565413
- [Background] Maagaard M, Heiberg J, Hjortdal VE. Small, unrepaired ventricular septal defects reveal poor exercise capacity compared with healthy peers: A prospective, cohort study. Int J Cardiol. 2017 Jan 15;227:631-634. doi: 10.1016/j.ijcard.2016.10.086. Epub 2016 Oct 29. PMID 27810297
- [Background] Maagaard M, Heiberg J, Asschenfeldt B, Ringgaard S, Hjortdal VE. Does functional capacity depend on the size of the shunt? A prospective, cohort study of adults with small, unrepaired ventricular septal defects. Eur J Cardiothorac Surg. 2017 Apr 1;51(4):722-727. doi: 10.1093/ejcts/ezw420. PMID 28204298
- [Background] Heiberg J, Petersen AK, Laustsen S, Hjortdal VE. Abnormal ventilatory response to exercise in young adults operated for ventricular septal defect in early childhood: A long-term follow-up. Int J Cardiol. 2015 Sep 1;194:2-6. doi: 10.1016/j.ijcard.2015.05.071. Epub 2015 May 15. PMID 26011258
- [Background] Rex CE, Eckerstrom F, Heiberg J, Maagaard M, Rubak S, Redington A, Hjortdal VE. Surgical closure of a ventricular septal defect in early childhood leads to altered pulmonary function in adulthood: A long-term follow-up. Int J Cardiol. 2019 Jan 1;274:100-105. doi: 10.1016/j.ijcard.2018.06.109. Epub 2018 Jul 2. PMID 30001944
- [Background] Gabriels C, De Backer J, Pasquet A, Paelinck BP, Morissens M, Helsen F, Van De Bruaene A, Budts W. Long-Term Outcome of Patients with Perimembranous Ventricular Septal Defect: Results from the Belgian Registry on Adult Congenital Heart Disease. Cardiology. 2017;136(3):147-155. doi: 10.1159/000448513. Epub 2016 Sep 21. PMID 27648950
- [Background] Asschenfeldt B, Heiberg J, Ringgaard S, Maagaard M, Redington A, Hjortdal VE. Impaired cardiac output during exercise in adults operated for ventricular septal defect in childhood: a hitherto unrecognised pathophysiological response. Cardiol Young. 2017 Oct;27(8):1591-1598. doi: 10.1017/S1047951117000877. Epub 2017 May 25. PMID 28539128
- [Background] Karonis T, Scognamiglio G, Babu-Narayan SV, Montanaro C, Uebing A, Diller GP, Alonso-Gonzalez R, Swan L, Dimopoulos K, Gatzoulis MA, Li W. Clinical course and potential complications of small ventricular septal defects in adulthood: Late development of left ventricular dysfunction justifies lifelong care. Int J Cardiol. 2016 Apr 1;208:102-6. doi: 10.1016/j.ijcard.2016.01.208. Epub 2016 Jan 23. PMID 26844920
- [Background] Shrout PE, Fleiss JL. Intraclass correlations: uses in assessing rater reliability. Psychol Bull. 1979 Mar;86(2):420-8. doi: 10.1037//0033-2909.86.2.420. PMID 18839484
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] DUBOIS AB, BOTELHO SY, BEDELL GN, MARSHALL R, COMROE JH Jr. A rapid plethysmographic method for measuring thoracic gas volume: a comparison with a nitrogen washout method for measuring functional residual capacity in normal subjects. J Clin Invest. 1956 Mar;35(3):322-6. doi: 10.1172/JCI103281. No abstract available. PMID 13295396
- [Background] Horsley A. Lung clearance index in the assessment of airways disease. Respir Med. 2009 Jun;103(6):793-9. doi: 10.1016/j.rmed.2009.01.025. Epub 2009 Feb 25. PMID 19246184
- [Background] Horsley AR, Gustafsson PM, Macleod KA, Saunders C, Greening AP, Porteous DJ, Davies JC, Cunningham S, Alton EW, Innes JA. Lung clearance index is a sensitive, repeatable and practical measure of airways disease in adults with cystic fibrosis. Thorax. 2008 Feb;63(2):135-40. doi: 10.1136/thx.2007.082628. Epub 2007 Aug 3. PMID 17675315
- [Background] Verbanck S, Thompson BR, Schuermans D, Kalsi H, Biddiscombe M, Stuart-Andrews C, Hanon S, Van Muylem A, Paiva M, Vincken W, Usmani O. Ventilation heterogeneity in the acinar and conductive zones of the normal ageing lung. Thorax. 2012 Sep;67(9):789-95. doi: 10.1136/thoraxjnl-2011-201484. Epub 2012 Apr 27. PMID 22544894
- [Background] Johnson DC. Importance of adjusting carbon monoxide diffusing capacity (DLCO) and carbon monoxide transfer coefficient (KCO) for alveolar volume. Respir Med. 2000 Jan;94(1):28-37. doi: 10.1053/rmed.1999.0740. PMID 10714476
- [Background] Shi Y, Aledia AS, Tatavoosian AV, Vijayalakshmi S, Galant SP, George SC. Relating small airways to asthma control by using impulse oscillometry in children. J Allergy Clin Immunol. 2012 Mar;129(3):671-8. doi: 10.1016/j.jaci.2011.11.002. Epub 2011 Dec 17. PMID 22178635
- [Background] Oostveen E, MacLeod D, Lorino H, Farre R, Hantos Z, Desager K, Marchal F; ERS Task Force on Respiratory Impedance Measurements. The forced oscillation technique in clinical practice: methodology, recommendations and future developments. Eur Respir J. 2003 Dec;22(6):1026-41. doi: 10.1183/09031936.03.00089403. PMID 14680096
- [Background] Beaver WL, Wasserman K, Whipp BJ. A new method for detecting anaerobic threshold by gas exchange. J Appl Physiol (1985). 1986 Jun;60(6):2020-7. doi: 10.1152/jappl.1986.60.6.2020. PMID 3087938
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Selskab DC. Anbefalinger for standardiseret minimumskrav til transthorakal ekkokardiografi hos voksne. In: Selskab DC, ed. Dansk Cardiologisk Selskab DCS: DCS, 2008.
- [Background] Brun H, Moller T, Fredriksen PM, Thaulow E, Pripp AH, Holmstrom H. Mechanisms of exercise-induced pulmonary hypertension in patients with cardiac septal defects. Pediatr Cardiol. 2012 Jun;33(5):782-90. doi: 10.1007/s00246-012-0216-9. Epub 2012 Mar 1. PMID 22383098
- [Background] Cheung MM, Smallhorn JF, McCrindle BW, Van Arsdell GS, Redington AN. Non-invasive assessment of ventricular force-frequency relations in the univentricular circulation by tissue Doppler echocardiography: a novel method of assessing myocardial performance in congenital heart disease. Heart. 2005 Oct;91(10):1338-42. doi: 10.1136/hrt.2004.048207. PMID 16162630
- [Derived] Maagaard M, Eckerstrom F, Schram AL, Jensen HAR, Hjortdal V. Health and Well-Being in Older Adults With a Surgically Closed or an Unrepaired Ventricular Septal Defect. J Am Heart Assoc. 2023 Aug 15;12(16):e028538. doi: 10.1161/JAHA.122.028538. Epub 2023 Aug 7. PMID 37548158
- [Derived] Eckerstrom F, Maagaard M, Boutrup N, Hjortdal VE. Pulmonary Function in Older Patients With Ventricular Septal Defect. Am J Cardiol. 2020 Jun 1;125(11):1710-1717. doi: 10.1016/j.amjcard.2020.02.014. Epub 2020 Mar 13. PMID 32291090